CLINICAL TRIAL: NCT04645927
Title: A Double-blinded, Randomized, Placebo-controlled Trial to Study the Effects of Dietary Flax Beverage on Memory and Cognition
Brief Title: Clinical Trial to Study the Effects of Dietary Flax Beverage on Memory and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Boniface Hospital (Other)
Collaborators: Pizzey Ingredients (Unknown); Canadian Agricultural Partnership (Unknown)
Responsible Party: Principal Investigator, Dr. Benedict C. Albensi, Principal Investigator and Professor, St. Boniface Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CT/2019/004
Record Dates: First submitted 2020-11-13; First posted 2020-11-27 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2023-08

CONDITIONS: Memory; Disturbance, Mild
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo control beverage group (Placebo Comparator): The placebo will be provided in the same unmarked plain packages and contain the same constituents, but without flax (control packages contain oat fiber and milk). For 180 days (6 months) participants will consume 2 servings of 330 ml of placebo beverage (i.e. normal fiber beverage; control) per day.
  Interventions: Dietary Supplement: control beverage
- Experimental flax beverage group (Experimental): Flax beverage (30 gr daily, oral) is presented in liquid form in plain unmarked packages. For 180 days (6 months) participants will consume 2 servings of 330 ml of flax beverage (treatment group; 30 gms flax/day beverage) per day.
  Interventions: Dietary Supplement: flaxseed beverage

INTERVENTIONS:
Dietary Supplement: flaxseed beverage — Pizzey Ingredients Inc. introduced a flax beverage product that is a plant-based beverage product that is designed as an alternative to non-diary "milks" (almond milk & soy milk). Each 330 ml serving of flax beverage contains 15 g flaxseed, which amounts to 3.75 gm of omega-3 fatty acid. Preventing MCI or even AD may be within reach, if appropriate measures are taken early enough using strategies such as dietary supplementation.
  Arms: Experimental flax beverage group
Dietary Supplement: control beverage — Oat fibre control. For 180 days (6 months) participants will consume 2 servings of 330 ml of placebo beverage (i.e. normal fiber beverage; control) per day.
  Arms: Placebo control beverage group

SUMMARY:
Investigate the effects of flax beverage consumption on memory and cognition in subjects with memory deficit (i.e., amnestic MCI). In addition, it will correlate PET scan results (for a limited number of participants) and blood biomarker data with memory test results.

DETAILED DESCRIPTION:
This study is a multisite, double-blinded, randomized, placebo-controlled trial to examine the effect of daily flax beverage consumption on memory and cognition. This trial will be conducted at the I.H. Asper Clinical Research Institute and at the John Buhler Research Centre, Health Sciences Centre in Winnipeg, Manitoba.

Sixty men and women diagnosed with mild cognitive impairment (MCI) aged 60 to 84 years will be recruited by using advertisements/flyers, radio/TV announcements, the Alzheimer's Society network and/or will be referred by a general practitioner. The participants will be randomly divided: 30 subjects in the flax-treatment group and 30 placed in the control - placebo group. For 180 days (6 months) participants will either consume 2 servings of 330 ml of flax beverage (treatment group; 30 gms flax/day beverage) or placebo beverage (i.e. normal fiber beverage; control) per day.

Potential candidates will first be screened in-person at the I.H. Asper Clinical Research Institute; the screening visit (SV1) will last about 2 hours. The subject will first be asked to read, understand and sign a consent form. Then they will be subject to a questionnaire, a medical history, a blood pressure (BP) measurement and 2 screening memory & cognition tests; Montreal Cognitive Assessment (MoCA), which is sensitive to MCI and the Depression Anxiety Stress Scale (DASS). Based on this initial in-person visit, investigators will determine participants' eligibility to continue in the study. Study staff will contact the Office of Clinical Research at St. Boniface Hospital to assign an eligible participant a unique study code.

If the participant meets the inclusion criteria based on their SV1 visit, investigators will plan a baseline visit for the participant. During the first baseline visit (BV1), if the subject is interested to take part in this study, they will be asked to perform the Cambridge Neuropsychological Test Automated Battery (CANTAB). This baseline visit will take about 1.0 hours to accomplish.

Investigators will then plan a second baseline visit (BV2) for a fasting blood draw, which will take approximately 15 minutes to complete. The participant will have to fast for 10 hours prior to their visit and a certified phlebotomist will collect approximately 16 mL of blood (about 3 teaspoons). In addition, investigators will review beverage consumption logs with participants and provide 30 days of beverage regime if they have a vehicle to take it home (if they have a car and are not scheduled for a PET scan).

A third baseline visit will be scheduled (BV3), where some participants will be randomly invited for a brain PET scan (10 controls from the placebo group and 10 from Flax-treatment group) at the baseline and at the end of the study. For this procedure the participant will need to fast for 4 hours. The participants have the option of declining the PET scans, if they wish.

The participants will need to be provided with 30 days of flax beverage every month (by either pickup or delivery). They also will need to submit their consumption log sheets (requested monthly) at this time to be reviewed by a study coordinator.

At the end of the study, the participants (T180) will have final follow up review of their medical history, blood pressure measurements and memory and cognitive tests (similar to those performed at the screening visit and baseline visit 1), along with a fasting blood draw (FV1, FV2). In addition, a third final study visit (FV3) will be scheduled for those who agreed to brain PET scans at the beginning of the study. In the final visit, an honorarium of $25.00 will be paid for their participation.

Each participant will visit the I.H Asper Clinical Research Institute a minimum of 5 times for the entire study. Those participants selected for brain PET scan will have 2 additional visits at John Buhler Research Centre, Health Sciences Centre; therefore, they will need a total of 7 visits for the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Normal thyroid function (as determined by case history).
* Patients must have MCI or Minor Neurocognitive Disorder according to DSM-5 (see definition of DSM-5 under List of Abbreviations on Page 5).
* Ability to provide written informed consent.
* Age 60 to 84.

Exclusion Criteria:

* Any diagnosis of Alzheimer's Disease (AD) or Dementia by a physician.
* MoCA Cognitive Test Score outside 19-25 inclusive (determined in first Baseline Visit).
* DASS Test Score: Severe or Extremely Severe Score for any of the 3 measurements (Depression, Anxiety or Stress) (determined in the first Baseline Visit).
* Allergies to any of the components of the Test Product or Placebo (see Section 7.5).
* Lactose Intolerance or Allergy to any of the product components.
* Vitamin E, Vitamin B (any form), fish oil, omega pills or flaxseed products.
* Any significant neurological disease as determined during screening (case history). Examples include Parkinson's, Huntington's, brain tumor, seizure disorders, subdural hematoma, multiple sclerosis, history of head trauma including multiple head trauma with loss of consciousness.
* Diagnosis of diabetes mellitus as determined during screening (case history).
* Significant cerebrovascular or cardiovascular disease as determined during screening (case history).
* Psychotic features or history of schizophrenia as determined during screening (case history).
* Another major psychiatric disorder as described in DSM 5 within the past 2 years (see definition of DSM 5 as described under List of Abbreviations on Page 5).
* History of alcohol or substance abuse as determined during screening (case history).
* History of systemic cancer as determined during screening (case history).
* Sudden changes in bowel movements for more than 2 weeks, undiagnosed rectal bleeding, or failure to defecate following the use of a laxative.
* Presence of abdominal pain, nausea, vomiting or fever.
* Difficulty in swallowing (dysphagia).
* Blood Pressure (systolic >180 and/or diastolic >110). A stable dose of hypertension drugs for elevated blood pressure during the course of the study is not exclusionary.
* Non AD Medications: Use of centrally active beta-blockers, narcotics, methyldopa and clonidine within 4 weeks prior to screening.
* Use of anti-Parkinsonian medications (e.g. Sinemet, amantadine, bromocriptine, pergolide & selegiline) within 2 months prior to screening.
* Use of neuroleptics or narcotic analgesics within 4 weeks prior to screening.
* Use of long-acting benzodiazepines or barbiturates within 4 weeks prior to screening.
* Use of short-acting anxiolytics or sedative hypnotics more frequently than 2 times per week within 4 weeks prior to screening (note: sedative agents should not be used within 72 hours of screening).
* Initiation or change in dose of an antidepressant lacking significant cholinergic side effects within the 4 weeks prior to screening (use of stable doses of antidepressants for at least 4 weeks prior to screening is acceptable).
* Use of systemic corticosteroids within 3 months prior to screening.
* Medications with significant cholinergic or anticholinergic side effects (e.g. pyridostigmine, tricyclic antidepressants, meclizine, and oxybutynin) within 4 weeks prior to screening.
* Use of anti-convulsants (e.g. Phenytoin, Phenobarbital, Carbamazepine) within 2 months prior to screening.
* Use of warfarin (Coumadin) within 4 weeks prior to screening.
* Any prior use of any FDA approved medications for the treatment of Alzheimer's disease (e.g. tacrine, donepezil, or other newly approved medications).
* Other: Subjects who, in the PI's opinion, will not comply with study procedures.

Ages: 60 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Cognitive/Memory score for CANTAB test. | About 1.0 hour to administer. The memory test will be administered two times, that is before and after flax beverage dietary supplementation that lasts for 6 months; which will occur at baseline (2nd visit) at then 6 months later.
  Cambridge Neuropsychological Test Automated Battery (CANTAB). CANTAB, a test to assess neurocognitive performance. There is no cut-off score for the CANTAB test and this test is non-exclusionary.

SECONDARY OUTCOMES:
Memory test using the Montreal cognitive assessment (MoCA) instrument | The test takes 15 mins. The test will be administered 2 times. First at the 1st visit or screening and then at the final visit 6 months later.
  MoCA is used as a screening tool to determine which participants are allowed to enter the trial. Participants will be included if their score ranges from 19-25 inclusive.
Depression Anxiety and Stress Scale (DASS) | The test takes 5 mins. Testing will be done at 2 time points, that is at the 1st screening visit and at 6 months.
  The DASS is a suitable instrument to screen for depressive disorders. A score of Severe or Extremely Severe for any of the 3 DASS measurements (Depression, Anxiety or Stress) will exclude the participant from the study.
Aberrant Brain PET scans. | One and one-half hours for each PET scan. The PET scans will be administered two times, which will occur at baseline (3rd visit) at then 6 months later.
  A subset of participants randomly selected will have a brain PET scan. Since a limited number of participants will have PET scan (10 flax beverage group, 10 control beverage group, n=20).
Blood draw. | Blood collection takes 5 minutes. Collection will take place at 2 time points, at a 3rd visit during baseline and at 6 months.
  Blood (16 ml) will be collected from each participant.
Blood pressure measurement. | Blood pressure measurements take 5 minutes. Blood pressure measurements will occur two times, which will occur at baseline - 2nd visit and then 6 months later.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Campbell, MD, Principal Investigator — St. Boniface Hospital
Locations (2):
- Canada (2):
  - I.H. Asper Clinical Research Institute, Winnipeg, Manitoba
  - Health Sciences Ctr., Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No